CLINICAL TRIAL: NCT03569397
Title: Music Therapy Versus Control During Total Knee Replacement Under Spinal Anesthesia
Brief Title: Music Therapy Versus Control for Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Promil Kukreja, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 56789012
Record Dates: First submitted 2018-06-15; First posted 2018-06-26 (Actual); Results first posted 2021-05-05 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2020-11

CONDITIONS: Arthroplasty, Replacement, Knee
MeSH Terms: interventions — Music Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music Therapy (Experimental): Administer music therapy during the operation
  Interventions: Other: Music Therapy
- Non-Music Therapy (No Intervention): No headphones or music therapy during the operation

INTERVENTIONS:
Other: Music Therapy — Patients will be administered music therapy during the operation.
  Arms: Music Therapy

SUMMARY:
For millennia, people have listened to and enjoyed music for entertainment, as a distraction from daily troubles, and as a means to relax and relieve stress. It is no real surprise that the relaxing and stress-relieving effects of music have been shown in patients having surgery. For patients having surgery with spinal anesthesia, music therapy during the operation decreases sedation requirements, anxiety and may improve patient satisfaction. Music therapy during surgery may also lead to a decreased stress response, as evidenced by more stable cortisol levels. Studies done previously have included patients undergoing various surgical procedures, however no studies have been done specifically for patients undergoing total knee arthroplasty. Because total knee arthroplasty is a common procedure usually done under spinal anesthesia at our institution, we would like to study the effects music therapy could have on our patient population.

DETAILED DESCRIPTION:
A. Patients who consent to the study will be randomized 1:1 to either the investigational group ("Music Therapy" group) or the control group ("No Music" group). Participants will be randomized using a random number generator.

B. Consent and study enrollment will occur in the preoperative area prior to surgery. After enrollment, all patients will complete a State-Trait Anxiety Assessment. Patients in the "Music Therapy" group will be asked to choose a genre of calming music that they would like to listen to during the operation (instrumental, jazz, classical). All patients enrolled in the study will continue to receive routine preoperative care but will also have a baseline cortisol level drawn. This blood draw will be compared to a cortisol level at the end of surgery to assess the patient's physiologic stress response to surgery.

a. After proceeding to the operating room, all patients will receive routine preoperative care during placement of spinal anesthesia. In addition to monitors routinely placed prior to spinal block, a Bi-Spectral Index monitor will be placed on the patient's forehead to monitor sedation levels during the procedure. A Bi-Spectral Index monitor is a noninvasive series of patches placed on the patient's forehead that, through a propriety equation creates a number (1-100) from processed electroencephalography waves that correlates with depth of sedation or anesthesia. After the spinal anesthetic block is placed, the patients in the "Music Therapy" group will wear headphones that will play their pre-selected music. The "No Music" group will receive intraoperative standard of care with no headphones. Headphones will be worn by the "Music Therapy" patients until the procedure is finished (skin incision is closed).

C. During the procedure, routine intraoperative sedation consisting of propofol, fentanyl and midazolam will be administered. All patients will be given 1 mg midazolam, 50 mcg fentanyl and propofol dosing titrated to maintain a Bi-Spectral Index level <70, which correlates to moderate sedation.9

D. At the end of the surgical procedure (within 30 minutes of incision closure), a serum cortisol level will be drawn to assess the physiologic stress response to surgery.

E. All patients will receive standard postoperative care in the post-anesthesia care.

F. On postoperative day 1, all patients will again complete a State-Trait Anxiety Assessment. Additionally, patients in the music therapy group will complete a satisfaction survey.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing total knee arthroplasty under spinal anesthesia.
* Patients 18 years of age or older.
* Patients classified by the American Society of Anesthesiology (ASA) class I, II, or III.

Exclusion Criteria:

* Any patient not classified as an ASA I, II, or III.
* Patients with hearing impairment, defined by personal endorsement of hearing impairment or use of hearing aids.
* Patients with contraindication to spinal anesthesia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2018-10-08 (Actual); Primary Completion 2019-12-18 (Actual); Study Completion 2020-03-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Promil Kukreja, MD, PhD, Principal Investigator — UAB Department of Anesthesiology
Locations (1):
- UAB Highlands Hospital, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kukreja P, Talbott K, MacBeth L, Ghanem E, Sturdivant AB, Woods A, Potter WA, Kalagara H. Effects of Music Therapy During Total Knee Arthroplasty Under Spinal Anesthesia: A Prospective Randomized Controlled Study. Cureus. 2020 Mar 24;12(3):e7396. doi: 10.7759/cureus.7396. PMID 32337122

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Music Therapy | Non-Music Therapy
Started | 29 | 28
Completed | 29 | 28
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Music Therapy | Non-Music Therapy | Total
Number analyzed (Participants) | 29 | 28 | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.14 (1.82) | 61.68 (2.27) | 62.3 (1.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 18 | 38
  Male | 9 | 10 | 19
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 29 | 28 | 57

OUTCOME MEASURES:

1. Primary Outcome: Patient Satisfaction
Description: On a scale of 1-5 (Likert scale) patients were asked to rank their satisfaction with their perioperative care. 1 indicates poor satisfaction, 5 indicates excellent satisfaction. Only patients in the music therapy group were asked for their satisfaction ranking.
Time Frame: Postoperative day 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Music Therapy
Number analyzed (Participants) | 29
score on a scale | 4.48 (0.16)

ADVERSE EVENTS:
Time Frame: From the time of discharge to 12 months post discharge
Arm/Group | Music Therapy | Non-Music Therapy
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/28
Other Adverse Events (participants affected / at risk) | 0/29 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-09): https://cdn.clinicaltrials.gov/large-docs/97/NCT03569397/Prot_SAP_000.pdf